CLINICAL TRIAL: NCT06958939
Title: A Single-center, Single-arm, Dose-exploration Study Evaluating the Safety and Efficacy of SENL103 Autologous T-cell Injection (S103) in the Treatment of Refractory Generalized Myasthenia Gravis
Brief Title: The Safety and Efficacy of S103 in the Treatment of Refractory Generalized Myasthenia Gravis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ting Chang, MD (Other)
Collaborators: Hebei Senlang Biotechnology Co., LTD (Unknown)
Responsible Party: Sponsor-Investigator, Ting Chang, MD, Associate Professor, Tang-Du Hospital
Organization: Tang-Du Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CART-20250321
Record Dates: First submitted 2025-04-13; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: Dose 1 1.0 × 10e6/kg S103 CAR-T cells
  Dose 2 2.0 × 10e6/kg S103 CAR-T cells
  Dose 3 4.0 × 10e6/kg S103 CAR-T cells
  Dose 4 8.0 × 10e6/kg S103 CAR-T cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S103 CAR-T (Experimental): This study adopted a single-arm design, with all patients receiving sequential administration of different doses of S103 CAR-T
  Interventions: Drug: Dose level 1 group; Drug: Dose level 2 group; Drug: Dose level 3 group; Drug: Dose level 4 group

INTERVENTIONS:
Drug: Dose level 1 group — 1.0 × 10e6/kg S103 CAR-T cells
Drug: Dose level 2 group — 2.0 × 10e6/kg S103 CAR-T cells
Drug: Dose level 3 group — 4.0 × 10e6/kg S103 CAR-T cells
Drug: Dose level 4 group — 8.0 × 10e6/kg S103 CAR-T cells

SUMMARY:
This study is a single-center, open-label, single-arm, dose-exploration study to evaluate the safety and preliminary effectiveness of BCMA CAR-T（S103） in the treatment of refractory, generalized myasthenia gravis. The study is a dose escalation trial in adult, refractory, systemic MG patients. A total of 6-24 MG patients who meet the inclusion criteria are expected to be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, ≤80 years;
2. MGFA classification type IIa-IVa;
3. Voluntary participation in the study: understanding and awareness of the study and voluntary signing of the informed consent form;
4. Meeting the diagnosis of myasthenia gravis;
5. Assessed by the investigator as meeting the diagnostic criteria for refractory MG: fulfilling one of the following 4 conditions:

   1. After adequate dose and duration of at least 2 conventional immunotherapies (including steroid and non-steroid immunosuppressants), the post-intervention status (PIS) is unchanged or worsened.
   2. After adequate dose and duration of at least 2 conventional immunotherapies, the PIS is improved, but the MG-ADL score remains

      * 6 for at least 6 months.
   3. After adequate dose and duration of at least 2 conventional immunotherapies, the PIS is remission or improvement, but during regular tapering of immunotherapy, there are still ≥2 exacerbations per year (MG-ADL score ≥6).
   4. The investigator considers that, despite current conventional immunotherapy, MG still imposes a significant functional burden on the patient.
6. MG-ADL score ≥6 or QMG score ≥11 at screening and baseline, with ocular muscle score less than 50% of the total score.

Exclusion Criteria:

1. Any medical or psychiatric condition that the investigator deems may endanger the study participant or affect their ability to participate in the study; or any condition the investigator considers associated with poor compliance;
2. Females who are breastfeeding or pregnant, or plan to become pregnant at any time during the 12-month period after receiving CAR-T therapy, or have a history of spontaneous or induced abortion within 4 weeks prior to screening;
3. Study participants with clinically relevant active infections (e.g., sepsis, pneumonia, or abscess) or severe infections (requiring hospitalization or antibiotic treatment) within 4 weeks prior to screening;
4. Thymectomy within 6 months prior to baseline or planned thymectomy during the study period, or thymoma requiring chemotherapy and/or radiotherapy at any time;
5. Study participants who received live attenuated vaccines within 8 weeks prior to screening; or plan to receive live vaccines within 8 weeks after treatment;
6. Study participants who received prior rituximab treatment within 6 months before screening;
7. Treatment with tocilizumab, eculizumab, or efgartigimod within 3 months prior to screening;
8. Intravenous immunoglobulin, plasma exchange, or immunotherapy within 4 weeks prior to screening;
9. Known severe underlying diseases, such as liver or kidney dysfunction, hematologic disorders, prior severe cardiovascular diseases, severe hypertension, diabetes, or poorly controlled blood pressure or blood glucose;
10. Unresected thymoma;
11. Rapid symptom deterioration during the lead-in period, progressing to crisis or pre-crisis state (MGFA IVb-V);
12. Other conditions deemed by the investigator as unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Day 28
  DLT is defined as the following conditions that occur during the DLT evaluation period, which are not attributed to disease progression or disease-related processes, but are related to the study drug:
  1. All treatments with grade 4 or 5 cytokine release syndrome (CRS);
  2. Grade ≥3 immune effector cell-associated neurotoxicity syndrome (ICANS) possibly related to CAR-T therapy in all treatments;
  3. Grade 3 hematologic toxicity lasting more than 7 days, not caused by the underlying disease (excluding lymphocyte count decrease due to lymphodepletion);
  4. Grade ≥3 organ toxicity reactions (cardiac, skin, gastrointestinal, hepatic, pulmonary, renal/genitourinary) possibly related to CAR-T therapy in all treatments, with cardiac toxicity and renal toxicity reactions ≥ grade 2 considered as DLT;
  5. Treatment-related death;
  6. Other toxicities determined to be DLT after discussion by the SRC.

SECONDARY OUTCOMES:
Proportion of subjects who reach MSE (ADL≤1 score, for 4 weeks) at 3 months and 6 months after infusion | 3 month, 6 month
  Myasthenia Gravis Activities of Daily Living (MG-ADL) is a questionnaire that includes 8 items: ptosis, diplopia, speech, chewing, swallowing, breathing, and upper and lower limb functions. The scale uses a 4-level scoring system, with a total score of 0-24, and higher scores indicate more severe disability, with an improvement of 2 points or more suggesting clinical improvement.
Changes in ADL score relative to baseline at 28 days, 3 months, 6 months after infusion | 28 days, 3 months, 6 months
  Myasthenia Gravis Activities of Daily Living (MG-ADL) is a questionnaire that includes 8 items: ptosis, diplopia, speech, chewing, swallowing, breathing, and upper and lower limb functions. The scale uses a 4-level scoring system, with a total score of 0-24, and higher scores indicate more severe disability, with an improvement of 2 points or more suggesting clinical improvement.
Changes in QMG score relative to baseline at 28 days, 3 months, 6 months after infusion | 28 days, 3 months, 6 months
  Quantitative Myasthenia Gravis scale(QMG), mainly measures the patient's muscle strength and endurance. The QMG assessment includes diplopia, ptosis, facial muscle strength, swallowing, articulation, arm lift on both sides, percentage of predicted forced vital capacity (FVC), head lift, grip strength on both hands, and leg lift on both sides in a supine position, with 13 items in total. Each item is scored from normal (0) to severe (3), with a total score ranging from 0 to 39, and a higher score indicates a more severe disease. A total score change of more than 3 points is considered clinically significant.
Changes in MGC score relative to baseline at 28 days, 3 months, 6 months after infusion | 28 days, 3 months, 6 months
  MG Composite (MG-C) combines physician-reported and patient-reported entries. The scale assesses 10 items, with talking, chewing, and swallowing indices self-assessed by study participants, with total scores ranging from 0 to 50. For most patients, a score change of ≥3 points is associated with clinically significant symptom change.
Changes in QOL15 score relative to baseline at 28 days, 3 months, 6 months after infusion | 28 days, 3 months, 6 months
  15-item MG-specific QOL scale, MG-QOL15, is a short survey questionnaire completed by participants, with 15 items covering three aspects: physical, psychological, and social. It aims to assess the "patient's perspective" of "quality of life" related to MG, using a 5-level scoring method (from mild to severe, 0-4 points), with a maximum score of 60 points, and higher scores indicating poorer quality of life.
Median time to re-infusion to achieve MSE status | 6 months
Changes of blood pressure | 28 days, 3 months, 6 months
Changes of pulse rate | 28 days, 3 months, 6 months
Changes of weight | 28 days, 3 months, 6 months
Changes in myasthenia gravis-specific autoantibody titers relative to baseline at 28 days, 3 months, 6 months after infusion | 28 days, 3 months, 6 months
Changes in immunoglobulins relative to baseline at 28 days, 3 months, 6 months after infusion | 28 days, 3 months, 6 months
Incidence and grading of severe adverse events (SAE) from 28 days to 2 years after re-infusion | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ting Chang, Study Chair — The Second Affiliated Hospital of Air Force Medical University
Locations (1):
- The Second Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Experimental data may be shared with the consent of the principal investigator
Supporting Information: ICF, CSR